CLINICAL TRIAL: NCT00142844
Title: Two Medications, Disulfiram and Naltrexone, in the Treatment of Patients With Both Cocaine and Alcohol Dependence
Brief Title: Combination of Disulfiram Plus Naltrexone to Treat Both Cocaine- and Alcohol-dependent Individuals - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Helen Pettinati, Ph.D., University of Pennsylvania Treatment Research Cener
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-12756-1; P50DA012756-01 (NIH); DPMC (Other: NIDA); NCT00136162 (obsolete NCT alias)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol-Related Disorders; Alcoholism; Cocaine-Related Disorders
Keywords: cocaine
MeSH Terms: conditions — Alcohol-Related Disorders; Alcoholism; Cocaine-Related Disorders | interventions — Naltrexone; Disulfiram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Naltrexone (Experimental): Naltrexone
  Interventions: Drug: Naltrexone
- Disulfiram (Experimental): Disulfiram
  Interventions: Drug: Disulfiram
- Naltrexone and Disulfiram (Experimental): Naltrexone and Disulfiram
  Interventions: Drug: Naltrexone; Drug: Disulfiram
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone
  Arms: Naltrexone; Naltrexone and Disulfiram
Drug: Disulfiram
  Arms: Disulfiram; Naltrexone and Disulfiram
Drug: Placebo
  Arms: Placebo

SUMMARY:
Many cocaine dependent individuals are also dependent on alcohol. Such individuals respond poorly to existing treatments and have received little research attention in the past. The purpose of this study is to determine whether the combination of naltrexone and disulfiram is useful in decreasing alcohol use and cravings in people diagnosed with both cocaine and alcohol dependence.

DETAILED DESCRIPTION:
Many cocaine dependent individuals are also dependent on alcohol. Such individuals respond poorly to existing treatments and have received little research attention in the past. Naltrexone and disulfiram are medications currently approved for treating alcohol dependence. These two medications have different mechanisms of action in the body. In combination they might be effective in treating individuals dually diagnosed with cocaine and alcohol dependence. The purpose of this study is to determine whether the combination of naltrexone and disulfiram is useful in decreasing alcohol cravings in individuals who are dependent on both cocaine and alcohol.

Participants in this 5-year, double-blind study will be randomly assigned to receive disulfiram, naltrexone, both, or placebo. Treatment will occur for a 3-month period, after which alcohol, cocaine use, and other biopsychosocial measures will be assessed at Months 6 and 9.

ELIGIBILITY:
Inclusion criteria:

* Meets DSM-IV criteria for both alcohol and cocaine dependence, as determined by the Structured Clinical Interview(SCID-IV)
* Successful completion of alcohol detoxification (i.e., 3 consecutive days of abstinence from alcohol)
* Use of at least $100 worth of cocaine in the 30 days prior to enrollment
* In the past 30 days, Subject used no less than $100 worth of cocaine and drank a minimum of 12 standard alcohol drinks/week (on average), having at least four days in 30 where at least four or more drinks were ingested, as determined by the Timeline Followback (TLFB) - adapted to collect daily cocaine use;
* Able to commute to the treatment research center
* Speaks, understands, and writes English
* Understands and signs the informed consent.

Exclusion Criteria:

* Abstinence from alcohol or cocaine for more than 30 days before signing consent form
* Current DSM-IV diagnosis of any psychoactive substance dependence other than Alcohol, Cocaine or Nicotine dependence, as determined by the SCID;
* Evidence of opiate use in the past 30 days as assessed by self-report and intake urine drug screen;
* History of unstable or serious medical illness, including need for opioid analgesics;
* Concomitant treatment with phenytoin or from same drug class, lithium, serotonin selective reuptake inhibitors, tricyclic antidepressants, MAOI's or narcotics; 6) Use of any investigational medication within the past 30 days;
* Severe physical or medical illness such as AIDS, active hepatitis or significant hepatocellular injury as evidenced by elevated bilirubin levels;
* Severe psychiatric symptoms, e.g., psychosis, suicidal or homicidal ideation or mania;
* Female patients who are pregnant, nursing, or not using a reliable method of contraception. Acceptable methods of birth control include: barrier (diaphragm or condom) with spermicide, intrauterine progesterone contraceptive system, levonorgestrel implant, medroxyprogesterone acetate contraceptive injection, oral contraceptives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 1999-09; Primary Completion 2005-03 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Amount of alcohol and drug use. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Helen M Pettinati, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Pettinati HM, Kampman KM, Lynch KG, Xie H, Dackis C, Rabinowitz AR, O'Brien CP. A double blind, placebo-controlled trial that combines disulfiram and naltrexone for treating co-occurring cocaine and alcohol dependence. Addict Behav. 2008 May;33(5):651-67. doi: 10.1016/j.addbeh.2007.11.011. Epub 2007 Nov 17. PMID 18079068
- See also: University of Pennsylvania Center for Studies of Addiction — http://www.med.upenn.edu/csa/